CLINICAL TRIAL: NCT04653363
Title: Evaluation of the Applicability and Reliability of the Three Meter Backwalk Test in Children With Cerebral Palsy (CP)
Status: Completed | Type: Observational
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hatice Adıgüzel, Principal Investigator, Kahramanmaras Sutcu Imam University
Other Study IDs: SankoUniv
Record Dates: First submitted 2020-11-26; First posted 2020-12-04 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-04

CONDITIONS: Cerebral Palsy; Cerebral Palsy Spastic Diplegia; Hemiplegic Cerebral Palsy; Gait, Hemiplegic; Gait, Spastic
Keywords: Cerebral Palsy; backward walk; reliability; gait
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: study1 is the patients who will be assessed by first rater.
  Interventions: Other: assessments
- 2: study2 is the patients who will be assessed by second rater.
  Interventions: Other: assessments
- 3: Theh are healty peers control patients who will be assessed by first rater.
  Interventions: Other: assessments

INTERVENTIONS:
Other: assessments — All assesments will be done by the first physiotherapist. But only 3m backward test will be done by the first and second physiotherapist in the first day and second day.
  Other Names: three meter backward test; Time Up and Go test; Timed Up and Down Stairs Test; Four Square Step Test; Functional Reach Test; Pediatric Berg Balance Scale; demografic information form; gross motor function classification system (GMFCS); modified ashworth scale; Communication Function Classification System

SUMMARY:
Cerebral palsy (CP) is a non-progressive disturbance in the development of movement and posture that occurs in the prenatal or postnatal period, causing activity limitations. Most children and adolescents with CP experience limitations in their walking skills. Restrictions in the walking ability of children with CP are an important issue for both parents and healthcare professionals involved in their treatment.

The evaluation of walking is of great importance in terms of determining the effectiveness of the physiotherapy program, shaping the program, planning orthopedic and surgical applications, and determining the effectiveness, especially in children with CP who have walking potential. In the literature, easy-to-use, valid and reliable observational gait analysis that can evaluate gait pathologies and clinical gait in children with CP are emphasized. These measurements are of great importance in clinical practice.The ability of backward walking gives the child a different task than normal, allowing the observation of body perception, trunk stability provided by anterior-posterior co-contractions, balance, correction and protective reactions.

DETAILED DESCRIPTION:
The main purpose of CP rehabilitation is to ensure that the child gains maximum functional independence by obtaining the optimal development potential. Therefore, walking restrictions are one of the important problems in children with CP.

The most common type in the CP classification is the spastic type. The types with the best functional independence level in this group are; hemiparetic and diparetic CP. They do not have a good motor coordination due to stability problems caused by deviations in the center during walking. This situation affects balance and walking performance. As children get older, impairments in their walking ability become more pronounced. In addition to all these problems, hypertonus, increased stretching reflex, muscle weakness, coactivation in antagonist muscles, posture disorders, loss of proprioception, muscle and joint deformities are other factors that cause gait disturbances in children with CP. Therefore, the walking problems of the child with CP should be examined more clearly. At this point, it assigns a different task to the child with the evaluation of backward walking, and provides observation of body perception, trunk stability provided by anterior-posterior co-contractions, balance, correction and protective reactions. This observation ensures that the problem that will guide the treatment is precisely determined.The only test that can be applied to evaluate the ability to walk back is the three meter backward walk test. This test has been found to be valid and reliable in both the elderly population and patients with total knee arthroplasty.In the literature, there is no study about the three-meter backwalk test in children with CP. In this study, it was aimed to evaluate the backward walking skills of children with CP with the three meter backward walk test and to examine the applicability and reliability of the three meter backward walk test in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-18 years with a diagnosis of Hemiparetic and Diparetic SP with a Gross Motor Function Classification System (GMFCS) Level ≤ 3
* Children diagnosed with CP with Communication Function Classification System (CFCS) ≤ 3
* Children with ≤ 3 according to the Modified Ashworth Scale (MASH)
* Complete range of passive range of motion in the ankle and knee joints
* Volunteering to participate in the study

Exclusion Criteria:

* Not having Botulinum toxin or surgical operation in the last 6 months
* Having contracture in the ankle and knee joints

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: - Children aged 8-18 years with a diagnosis of Hemiparetic and Diparetic SP with a Gross Motor Function Classification System (GMFCS) Level ≤ 3
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
three meter backward walk test | first evaulation of first day of assessment (observer1), second evaulation of first day of assessment (observer2), second evaulation of second day of assessment (observer1, second evaulation of second day of assessment (observer2)
  Three meters of distance will be measured and marked. When the signal is given, they will be asked to walk backwards safely and stop when they reach the marked point. Patients will be allowed to look back if they wish. The person conducting the test will walk with the patients for safety. The measurements will be repeated 3 times and the average of the times will be recorded.

SECONDARY OUTCOMES:
Timed Up and Go Test | first day of assessment
  TUG is a reliable test that measures walking speed, postural control, functional mobility, and balance. For TUG measurement, the child will be seated in a height-adjustable chair. The height of the seat will be adjusted so that the subject's knees and hips are bent up to 90 degrees while sitting with their feet. A distance of 3 meters will be marked. When the child is given a command, he will be asked to walk up to the marked area and return. In the meantime, times are recorded. In addition, the test will be repeated 3 times and the average time will be recorded.
Timed Up and Down Stairs Test | first day of assessment
  This test will be carried out on a ladder with 14 steps and a step height of 19.5 cm. While the use of shoes is permitted during the test, the use of orthoses will not be allowed. The child will start the test at a distance of 30 cm from the lowest step. It will be asked to go up and down again safely, the time will be recorded. In addition, the test will be repeated 3 times and the average time will be recorded.
Four Square Step Test | first day of assessment
  A square divided into 4 sections will be created on a flat floor. Squares will be numbered. The child will stand in square 1, facing square 2. He will be asked to move to the squares 2-3-4-1-4-3-2-1 respectively. Thus, the child will be able to move back and forth right and left. It will be said that both feet must touch the ground. The period will start with the contact of the foot on the number 2 square and end with the contact of the number 1 square. The test will be applied 2 times and the good time will be taken.
Functional Reach Test | first day of assessment
  The child will be asked to stand sideways on a wall and keep the elbows in extension at 90 degrees of shoulder flexion without touching the wall. The first measurement will be made at this position. He will then be asked to stretch forward without taking any steps. The last point it can reach will be recorded. These two distances will be measured and recorded in meters. The test will be repeated when stepping or the foot is cut off from the ground.
Pediatric Berg Balance Scale | first day of assessment
  Balance assessment of the children to be included in the study will be made with the Pediatric Berg Balance Scale. The scale consists of 14 parts and each part is scored between 0 and 4. The highest score that can be obtained from the scale is 56. In the PBRS, the sections in the standard BDI are listed from easy to difficult.

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıgüzel, PhD, Study Director — sanko Üniversitesi
Locations (2):
- Turkey (Türkiye) (2):
  - Hatice Adıgüzel, Gaziantep, Batıkent
  - Hatice Adıgüzel, Gaziantep

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Celik OF, Adiguzel H, Kirmaci ZIK, Erel S, Demirguc A. Validity and reliability of the 3-meter backward walk test in children with cerebral palsy. Acta Neurol Belg. 2023 Aug;123(4):1439-1446. doi: 10.1007/s13760-023-02259-1. Epub 2023 Apr 4. PMID 37014515